CLINICAL TRIAL: NCT02973646
Title: Investigation on Antiviral Therapy of Peginterferon Alfa-2b in HBeAg Positive Chronic Hepatitis B Patients Based on Detection of Interferon Gene Mutation and Interferon Receptor
Brief Title: Peginterferon Alfa-2b Treatment in HBeAg(+) Chronic Hepatitis b Patients Based on Interferon Gene Mutation and Receptor Detection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Associated Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL2
Record Dates: First submitted 2016-11-13; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis b; peginterferon alfa-2b; interferon gene mutation; interferon receptor
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nucleos(t)ide analogues treatment (Experimental): Patients with interferon receptor level down-regulated at the 24th week. Patients of this group will receive peginterferon alfa-2b injection 80ug/d from baseline to 24th week, then nucleos(t)ide analogues (entecavir tablet 0.5mg/d or tenofovir tablet 300mg/d) from 25th to 36th week, then peginterferon alfa-2b injection 80ug/d again from 36th to 48th week.
  Interventions: Drug: Entecavir or Tenofovir; Drug: Peginterferon Alfa-2B
- Peginterferon treatment (Active Comparator): Patients with interferon receptor level not down-regulated at the 24th week. Patients of this group will receive peginterferon alfa-2b injection 80ug/d from baseline to 48th week.
  Interventions: Drug: Peginterferon Alfa-2B

INTERVENTIONS:
Drug: Entecavir or Tenofovir — Patients in nucleos(t)ide analogues treatment for 12 weeks group will receive nucleos(t)ide analogs therapy (Entecavir tablet 0.5mg/d or Tenofovir tablet 300mg/d) from Week 25th to 36th.
  Other Names: Baraclude; Viread
  Arms: Nucleos(t)ide analogues treatment
Drug: Peginterferon Alfa-2B

SUMMARY:
The study is to observe the anti-HBV therapeutic effects of peginterferon alfa-2b in chronic hepatitis b patients with e antigen positive based on the detection of interferon gene mutation (IFNA2 p.Ala120Thr) and interferon receptor (IFNAR2) detection.

DETAILED DESCRIPTION:
Patients with e antigen positive chronic hepatitis b were enrolled in the study. Age, sex, symptoms (e.g., fever, fatigue, poor appetite, jaundice) were recorded in the study. We also observed the laboratory test results including the levels of white blood cells (WBC), red blood cells (RBC), hemoglobin (HGB), platelet (PLT), alanine transaminase (ALT), aspartate transaminase (AST), hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis B e antibody (HBeAb), and hepatitis B virus (HBV) DNA; detection of gene mutation (IFNA2 p.Ala120Thr), levels of interferon receptor (IFNAR2).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis b Patients who should receive anti-HBV therapy according to guideline and are willing to receive interferon therapy;
2. Hepatitis B e antigen positive.

Exclusion Criteria:

1. Patients received anti-HBV therapy in the past 6 months;
2. Patients with liver cirrhosis or hepatocellular carcinoma or other malignancies;
3. Patients with other factors causing active liver diseases;
4. Pregnancy or lactation women;
5. Patients with HIV infection or congenital immune deficiency diseases;
6. Patients with severe diabetes, autoimmune diseases, other important organ dysfunctions and other serious complications.
7. Patients with other reasons not suitable to receive interferon therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
good virologic response | 24th week
  level of HBsAg is less than or equal to 1500 IU/ml

SECONDARY OUTCOMES:
common virologic response | 24th week
  level of HBsAg is more than 1500 IU/ml, also less than or equal to 20000 IU/ml
bad virologic response | 24th week
  level of HBsAg is more than 20000 IU/ml, level of HBV DNA is equal to or more than 4.0 log10 IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China